CLINICAL TRIAL: NCT01320826
Title: Prospective Study of the Quality of Colonoscopies Performed by Primary Care Endoscopists in Alberta, Canada
Brief Title: The Alberta Primary Care Endoscopy (APC-Endo) Study
Acronym: APC-Endo
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Alberta Ministry of Health - Alberta Rural Physician Action Plan (Unknown)
Responsible Party: Principal Investigator, Brian Rowe, Associate Dean (Clinical Research), Faculty of Medicine and Dentistry Canada Research Chair in Emergency Airway Diseases Professor and Research Director Department of Emergency Medicine, University of Alberta, University of Alberta
Other Study IDs: 2011-APCEndo-MK
Record Dates: First submitted 2011-03-03; First posted 2011-03-23 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Screening Test; Endoscopy; Colon Disease
Keywords: colonoscopy; primary care physicians; quality assurance
MeSH Terms: conditions — Colonic Diseases | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physician colonoscopists: All primary care physicians (family physicians and general internists) who perform colonoscopies were approached to voluntarily participate in the APC-Endo study.
  All patients having a colonoscopy done by an APC-Endo study physician endoscopist were approached at the time of their endoscopy to consent to the post procedure telephone survey.
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — Data pertaining to all colonoscopies performed by a APC-Endo study physician over a two month period will be collected.

SUMMARY:
It is hypothesized that primary care colonoscopists are able to achieve benchmarks in colonoscopy quality including cecal intubation and adenoma detection rates and serious adverse event rates.

This prospective study is the first in depth analysis of the quality of colonoscopic procedures performed by primary care physicians at a provincial level in Canada.

In addition, the APC Endo study is the first to directly examine both the quality of colonoscopy and patient satisfaction in the same study.

DETAILED DESCRIPTION:
Discrepant data exists about the quality of colonoscopies performed by family physicians and general internists. Currently in Canada, gastroenterologists and general surgeons perform 97% of the colonoscopies, but excessive wait times highlight a shortage of colonoscopists in Canada. This shortage will invariably worsen as our population ages and more Canadians become screened for colorectal cancer.

One method of improving this relative shortage of colonoscopists is through training primary care physicians in GI medicine and endoscopy. In order these physicians to be a legitimate option in the provision of colonoscopies; however, it must be shown that, as a group, they are able to meet benchmarks in colonoscopy competency.

This multi-centre observational study will be the first study to prospectively analyze colonoscopic examinations performed by primary care physicians at a provincial level. Using primarily cecal intubation rates and adenoma detection rates, along with other quality parameters, this study will compare the results of Alberta primary care physicians to standard benchmarks in colonoscopy competency.

Data will be collected using case report forms completed at the time of the colonoscopy, reviewing the patients' colonoscopy pathology results and a post procedure telephone survey to examine patient satisfaction rates.

If this study demonstrates that quality benchmarks are indeed met, then future training of primary care physicians in gastrointestinal medicine and endoscopy would be encouraged to help address current and future colonoscopist shortages.

ELIGIBILITY:
Inclusion Criteria:

* All patients having a colonoscopy done by an APC-Endo physician endoscopist during the study period will be approached at the time of their endoscopy to consent to the post procedure telephone.

Exclusion Criteria:

* Patients under the age of 18 years old
* Patients who will be unable to be contacted for the post procedure telephone survey. (e.g., moving out of the country in the following month)
* Patients who are unable to understand or speak basic English
* Patients who are cognitively impaired such that they were not able to complete the initial consent for their colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physician colonoscopists: All Albertan family physicians and general internists who perform colonoscopies will be invited to voluntarily participate in anonymized data collection pertaining to the quality of colonoscopies they perform over a two month period.
  All patients having a colonoscopy done by an APC-Endo physician endoscopist during the study period will be approached at the time of their endoscopy to consent to the post procedure telephone survey.
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Kolber, MD, CCFP, Study Director — University of Alberta; Brian H Rowe, MD, CCFP(EM), Principal Investigator — University of Alberta
Locations (13):
- Canada (13):
  - Barrhead Healthcare Centre, Barrhead, Alberta
  - Bonnyville Healthcare Centre, Bonnyville, Alberta
  - St. Mary's Hospital, Camrose, Alberta
  - Daysland Health Centre, Daysland, Alberta
  - Queen Elizabeth 2 Hospital, Grande Prairie, Alberta
  - William J. Cadzow Health Centre, Lac La Biche, Alberta
  - Sacred Heart Hospital, McLennan, Alberta
  - Peace River Community Health Centre, Peace River, Alberta
  - Pincher Creek Hospital, Pincher Creek, Alberta
  - Ponoka Hospital and Care Centre, Ponoka, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta
  - Taber Hospital, Taber, Alberta
  - Whitecourt Healthcare Centre, Whitecourt, Alberta

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled if they were undergoing a colonoscopy for any reason with one of the participating study primary care colonoscopists. Due to staggered local study start dates, data collection occurred between March 15, 2010 and June 14, 2010 and patient satisfaction phone surveys were completed by August 2010.
Groups:
- Patients Undergoing Colonoscopy: All patients having a colonoscopy done by an APC-Endo study physician endoscopist were approached at the time of their endoscopy to consent to the post procedure telephone survey.
Period: Overall Study
Arm/Group | Patients Undergoing Colonoscopy
Started | 577
Completed | 577
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants.: All patients having a colonoscopy done by an APC-Endo study physician endoscopist were approached at the time of their endoscopy to consent to the post procedure telephone survey.
Arm/Group | Participants.
Number analyzed (Participants) | 577
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 415
  >=65 years | 162
Age Continuous [Mean (Standard Deviation); unit: years] | 57.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295
  Male | 282
Region of Enrollment [Number; unit: participants]
  Canada | 577

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful Cecal Intubations (Crude)
Description: The percentage of successful cecal intubations (crude) = (total # of colonoscopies performed where cecal intubation was achieved / total # of colonoscopies attempted) x 100
Time Frame: At time of colonoscopy (DAY 1 of study)
Population: Prospective, observational study, all study participants were analyzed
Measure: Number (95% Confidence Interval); unit: percentage of colonoscopies performed
Groups:
- Percentage of Successful Cecal Intubations (Crude): The percentage of successful cecal intubations (crude) = (total # of colonoscopies performed where cecal intubation was achieved / total # of colonoscopies attempted) x 100
Arm/Group | Percentage of Successful Cecal Intubations (Crude)
Number analyzed (Participants) | 577
percentage of colonoscopies performed | 95.3 [93.3 to 96.9]

2. Primary Outcome: Percentage of Successful Cecal Intubations (Adjusted)
Description: The percentage of successful cecal intubations (adjusted) = total number of colonoscopies performed where cecal intubation was achieved / (total number of colonoscopies attempted -incomplete colonoscopies due to poor bowel preparation, colonic stricture, equipment failure or severe endoscopic colitis)
Time Frame: At time of colonoscopy (DAY 1 of study)
Measure: Number (95% Confidence Interval); unit: percentage of colonoscopies attempted
Groups:
- Percentage of Successful Cecal Intubations: The percentage of successful cecal intubations (adjusted) = total number of colonoscopies performed where cecal intubation was achieved / (total number of colonoscopies attempted -incomplete colonoscopies due to poor bowel preparation, colonic stricture, equipment failure or severe endoscopic colitis)
Arm/Group | Percentage of Successful Cecal Intubations
Number analyzed (Participants) | 577
percentage of colonoscopies attempted | 96.5 [94.6 to 97.8]

3. Primary Outcome: Adenoma Detection Ratio
Description: The adenoma detection ratio is the number of pathologically verified adenomas per number of colonoscopies performed. Adenoma detection ratio = total number of pathologically confirmed adenomas / number of colonoscopies attempted.
Time Frame: When pathology from colonoscopy available (on average 2-3 weeks after procedure)
Population: Number of patients who underwent colonoscopy
Measure: Number (95% Confidence Interval); unit: adenomas / colonoscopy
Groups:
- Adenoma Detection Ratio: The adenoma detection ratio is the number of pathologically verified adenomas per number of colonoscopies performed. Adenoma detection ratio = total number of pathologically confirmed adenomas / number of colonoscopies attempted.
Arm/Group | Adenoma Detection Ratio
Number analyzed (Participants) | 577
adenomas / colonoscopy | 0.62 [0.51 to 0.74]

4. Primary Outcome: Percentage of Males 50 Years and Older Undergoing First Time Colonoscopy With an Adenoma
Description: Percentage of patients with an adenoma = (number of patients who had at least one adenoma detected on colonoscopy / total number of colonoscopies attempted) x 100.
  For this specific outcome: we explored this outcome for males 50 years and older undergoing first time colonoscopy.
Time Frame: When pathology from colonoscopy available (on average 2-3 weeks after procedure)
Population: We only examined this outcome for males 50 years and older having their first colonoscopy
Measure: Mean (95% Confidence Interval); unit: percentage of males
Groups:
- Percentage of Males 50 Years and Older Undergoing First Time c: Percentage of patients with an adenoma = (number of patients who had at least one adenoma detected on colonoscopy / total number of colonoscopies attempted) x 100.
  For this specific outcome: we explored this outcome for males 50 years and older undergoing first time colonoscopy.
Arm/Group | Percentage of Males 50 Years and Older Undergoing First Time c
Number analyzed (Participants) | 282
percentage of males | 46.4 [38.5 to 54.3]

5. Secondary Outcome: Colonoscopy Complications: Bleeding, Perforation, Cardiopulmonary Complications Secondary to Conscious Sedation, and Death.
Description: Potential serious complications of colonoscopy include bleeding, perforation, cardiopulmonary complications secondary to conscious sedation and death.
  Potential serious complications will be determined from the case report form (physician reported) and at patient satisfaction phone survey (on average four weeks after colonoscopy).
  All potential serious complications of colonoscopy will be externally adjudicated.
Time Frame: Within four (4) weeks of colonoscopy
Measure: Number; unit: patients undergoing colonoscopy
Groups:
- Colonoscopy Complications: Potential serious complications of colonoscopy include bleeding, perforation, cardiopulmonary complications secondary to conscious sedation and death.
  Potential serious complications will be determined from the case report form (physician reported) and at patient satisfaction phone survey (on average four weeks after colonoscopy).
  All potential serious complications of colonoscopy will be externally adjudicated.
Arm/Group | Colonoscopy Complications
Number analyzed (Participants) | 577
patients undergoing colonoscopy | 4

6. Secondary Outcome: Colonoscopy Withdraw Time in Cases Where no Lesions Found
Description: Withdrawal time will be defined as the time from leaving the cecum until the colonoscope exits the anus. This will be calculated for cases in which no lesions were found.
Time Frame: At time of colonoscopy (DAY 1 of study)
Population: Only examined patients in which no lesions were detected.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Withdraw Times, Minutes
Number analyzed (Participants) | 295
minutes | 7 [6.6 to 7.4]

7. Secondary Outcome: Patient Comfort During Colonoscopy
Description: To determine the patients' comfort level during the colonoscopy, a five-item question used by the Joint Advisory Group on Gastrointestinal Endoscopy in the United Kingdom will be used.
  Patient discomfort on the 5 point scale:
  0 is no discomfort;
  1. is one or two episodes of discomfort, well tolerated;
  2. is more than two episodes of discomfort adequately tolerated;
  3. is significant discomfort experienced several times during the procedure;
  4. is extreme discomfort experienced frequency throughout the procedure.
  Minimum value = 0, maximum value = 4 with 4 being worse.
Time Frame: At time of colonoscopy (DAY 1 of study)
Measure: Mean (Standard Deviation); unit: units on the scale
Groups:
- Patient Comfort During Colonoscopy: Patient discomfort on 5 point scale 0 is no discomfort; 1 is one or two episodes of discomfort, well tolerated; 2 is more than two episodes of discomfort adequately tolerated; 3 is significant discomfort experienced several times during the procedure; 4 is extreme discomfort experienced frequency throughout the procedure.
Arm/Group | Patient Comfort During Colonoscopy
Number analyzed (Participants) | 577
units on the scale | 0.8 (0.79)

8. Secondary Outcome: Patient Satisfaction With Endoscopy Wait Time
Description: Patient satisfaction with endoscopy wait time will be recorded using a 7 point Likert scale at the time of the patient phone survey. 7 is extremely satisfied and 1 is extremely dissatisfied
  minimum score = 1 maximum score = 7
Time Frame: At patient satisfaction phone survey (on average 4 weeks after colonoscopy)
Population: 443 patients completed the post procedural satisfaction survey.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Patient Wait Time Satisfaction: Patient satisfaction with endoscopy wait time will be recorded using a 7 point Likert scale at the time of the patient phone survey. 7 is extremely satisfied and 1 is extremely dissatisfied
  minimum score = 1 maximum score = 7
Arm/Group | Patient Wait Time Satisfaction
Number analyzed (Participants) | 443
units on a scale | 7 [5 to 7]

9. Secondary Outcome: Patient Satisfaction With Hospital Experience for Colonoscopy
Description: Patient satisfaction with their hospital experience during their colonoscopy will be recorded by using a 7 point Likert scale at the time of the patient satisfaction phone survey.
  7 = extremely satisfied
  1 = extremely dissatisfied
  Minimum score = 1 Maximum score = 7
Time Frame: At patient satisfaction phone survey (on average 4 weeks after colonoscopy)
Population: 443 patients consented to and completed the post procedural satisfaction survey.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Patient Satisfaction With Hospital Experience: Patient satisfaction with hospital experience measured on 7 point Likert scale. 7 is extremely satisfied, 1 is extremely dissatisfied.
Arm/Group | Patient Satisfaction With Hospital Experience
Number analyzed (Participants) | 443
units on a scale | 7 [6 to 7]

10. Secondary Outcome: Colonoscopy Procedure Time
Description: Colonoscopic procedural time will be defined as the time from the first insertion of the colonoscope until it is removed from the anus.
Time Frame: At time of colonoscopy (DAY 1 of study)
Measure: Mean (95% Confidence Interval); unit: minutes
Groups:
- Procedural Time: Procedural time was defined as the time from the first insertion of the colonoscope until it was removed from the anus, in minutes
Arm/Group | Procedural Time
Number analyzed (Participants) | 577
minutes | 23.6 [22.7 to 24.5]

11. Secondary Outcome: Percentage of Patients Referred to a Specialist.
Description: The percentage of patients who are anticipated to be referred to specialists, for the gastrointestinal complaint for which the colonoscopy was performed will be determined and the reason for referral will be tabulated. The referral percentage will be determined both from the time of colonoscopy (physician reported) and from the patient satisfaction phone survey (patient reported).
Time Frame: Within four (4) weeks of colonoscopy
Measure: Number; unit: percentage of patients
Groups:
- Percentage of Patients Referred to a Specialist.: The percentage of patients who, after having a colonoscopy, are referred to another specialist for their gastrointestinal problem. A specialist was defined as a physician more specialized than the person performing the colonoscopy, and a referral was counted if the physician, at the time of colonoscopy, sent or anticipated sending the patient to a specialist for any reason, or if the patient believed they were being sent to a specialist.
Arm/Group | Percentage of Patients Referred to a Specialist.
Number analyzed (Participants) | 577
percentage of patients | 4.8

12. Primary Outcome: Percentage of Females 50 Years and Older Undergoing First Time Colonoscopy With an Adenoma
Description: Percentage of patients with an adenoma = (number of patients who had at least one adenoma detected on colonoscopy / total number of colonoscopies attempted) x 100.
  For this specific outcome: we explored this outcome for females 50 years and older undergoing first time colonoscopy.
Time Frame: [When pathology from colonoscopy available (on average 2-3 weeks after procedure)]
Population: For this outcome, we only examined females ≥ 50 years old having their first colonoscopy
Measure: Mean (95% Confidence Interval); unit: percentage of females
Groups:
- Percentage of Females ≥ 50 Years With an Adenoma: Percentage of patients with an adenoma = (number of patients who had at least one adenoma detected on colonoscopy / total number of colonoscopies attempted) x 100.
  For this specific outcome: we explored this outcome for females 50 years and older undergoing first time colonoscopy.
Arm/Group | Percentage of Females ≥ 50 Years With an Adenoma
Number analyzed (Participants) | 295
percentage of females | 30.2 [22.3 to 38.2]

ADVERSE EVENTS:
Arm/Group | Participants.
Serious Adverse Events (participants affected / at risk) | 4/577
Other Adverse Events (participants affected / at risk) | 0/577
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants. (N=577)
Perforation (Gastrointestinal disorders) | 1 (1)
Bleeding (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No